CLINICAL TRIAL: NCT06569511
Title: Predictive Value of NT-proBNP on Major Adverse Cardiovascular Events in Patients With Acute Coronary Syndrome During a 6-month Follow-up
Brief Title: Predictive Value of NT-proBNP on MACEs After Acute Coronary Syndrome
Acronym: MACEstdy
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Az, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: 164-2023
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Acute Coronary Syndrome; ST-segment Elevation Myocardial Infarction (STEMI); Non-ST-Segment Elevation Myocardial Infarction (NSTEMI); Major Adverse Cardiac Events
Keywords: NT-proBNP; MACEs; Acute coronary syndrome; STEMI; NSTEMI
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In patients diagnosed with Acute Coronary Syndrome based on anamnesis, clinical findings, electrocardiogram (ECG), and/or serum high-sensitivity cardiac troponin (hs-cTn) level in the Emergency Department, blood samples for serum N-terminal pro-B-type natriuretic peptide (NT-proBNP) value was additionally taken during transfer to the coronary intensive care unit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MACE-positive: Patients who have experienced a major adverse cardiovascular event (MACE) within a 6-month period after percutaneous coronary intervention (PCI), including nonfatal ischemic stroke, nonfatal myocardial infarction, cardiovascular mortality, or emergency department admission due to heart failure.
  Interventions: Diagnostic Test: N-terminal pro-B-type natriuretic peptide (NT-proBNP); Diagnostic Test: high sensitive cardiac troponin T (hs-cTnT)
- MACE-negative: Patients who have not experienced a major adverse cardiovascular event (MACE) within a 6-month period after percutaneous coronary intervention (PCI), including nonfatal ischemic stroke, nonfatal myocardial infarction, cardiovascular mortality, or emergency department admission due to heart failure.
  Interventions: Diagnostic Test: N-terminal pro-B-type natriuretic peptide (NT-proBNP); Diagnostic Test: high sensitive cardiac troponin T (hs-cTnT)

INTERVENTIONS:
Diagnostic Test: N-terminal pro-B-type natriuretic peptide (NT-proBNP) — In patients diagnosed with Acute coronary syndrome, blood samples for serum NT-proBNP value were taken during transfer to the coronary intensive care unit
Diagnostic Test: high sensitive cardiac troponin T (hs-cTnT) — In patients diagnosed with Acute coronary syndrome, serum high-sensitive cardiac troponin T (hs-cTnT) levels were measured on admission to the Emergency Department.

SUMMARY:
The role of N-terminal pro-B-type natriuretic peptide (NT-proBNP) as a cardiac biomarker in predicting short-term major adverse cardiovascular events (MACEs) in patients with Acute coronary syndrome (ACS) has been insufficiently reported and remains poorly understood. Additionally, the relationship between NT-proBNP levels and specific ACS subtypes has not been thoroughly examined. Therefore, our study investigated the predictive value of high-sensitivity cardiac troponin (hs-cTn) and NT-proBNP levels on admission for 6-month MACEs in patients who presented to the emergency department (ED) with ACS and subsequently underwent percutaneous coronary intervention (PCI). Furthermore, we sought to evaluate the association between MACEs and specific ACS subtypes.

DETAILED DESCRIPTION:
In patients diagnosed with Acute coronary syndrome (ACS) based on anamnesis, clinical findings, electrocardiogram (ECG), and/or serum high-sensitivity cardiac troponin (hs-cTn) level in the emergency department (ED), blood samples for serum N-terminal pro-B-type natriuretic peptide (NT-proBNP) value was additionally taken during transfer to the coronary intensive care unit, and left ventricular ejection fraction (LVEF) was calculated by echocardiography before percutaneous coronary intervention (PCI). In addition, demographics (age, sex, and smoking status), comorbidities (hypertension, diabetes mellitus [DM] and/or coronary artery disease [CAD]), initial complaints and diagnoses, vital signs (systolic blood pressure [SBP], heart rate [HR], and peripheral capillary oxygen saturation [SpO2]), laboratory parameters (serum creatinine, C-reactive protein, and hs-cTn), and ACS subtypes (ST-elevation Myocardial infarction [STEMI], non-ST-elevation Myocardial infarction [NSTEMI], or unstable angina pectoris [USAP]) were obtained during admission. GRACE risk score was calculated for each patient on admission using eight variables, including age, SBP, HR, and serum creatinine. At the end of the 6-month follow-up period, LVEF of surviving patients was assessed by control echocardiography. The short-term MACEs (e.g., nonfatal ischemic stroke, nonfatal myocardial infarction, cardiovascular mortality, or ED admission due to heart failure) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) who were admitted to the emergency department with Acute coronary syndrome and underwent percutaneous coronary intervention between September 2023 and February 2024.

Exclusion Criteria:

* patients younger than 18 years
* patients had no vascular lesions detected on percutaneous coronary intervention,
* patients had infective or structural cardiac pathologies (myocarditis, pericarditis, hypertrophic or dilated cardiomyopathies)
* patients had chronic heart failure with LVEF <40%, class 3 and 4 in the Killip classification
* patients had a diagnosis of malignancy, chronic renal failure, chronic liver failure, and a history of multiple trauma or surgery within the last month

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This prospective, observational, and single-center study included a total of 241 consecutive adult patients (≥18 years old) who were admitted to the emergency department with Acute coronary syndrome, including ST-elevated myocardial infarction, non-ST-elevated myocardial infarction, or Unstable Angina Pectoris between September 2023 and February 2024.
Sampling Method: Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Predictive ability of NT-proBNP for 6-months MACEs | From admission to 6 months
  The investigators assessed the effectiveness of N-terminal pro-B-type natriuretic peptide (NT-proBNP) value at admission in predicting 6-months major adverse cardiovascular events (MACEs) in patients with acute coronary syndrome.

SECONDARY OUTCOMES:
Incidence of MACEs in STEMI | From admission to 6 months
  The investigators assessed the incidence of major adverse cardiovascular events (MACEs) in patients with ST-elevation myocardial infarction (STEMI).
Incidence of MACEs in NSTEMI | From admission to 6 months
  The investigators assessed the incidence of major adverse cardiovascular events (MACEs) in patients with non-ST-elevation myocardial infarction (NSTEMI).
Incidence of MACEs in USAP | From admission to 6 months
  The investigators assessed the incidence of major adverse cardiovascular events (MACEs) in patients with unstable angina pectoris (USAP).

CONTACTS AND LOCATIONS:
Overall Officials: Adem Az, M.D., Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Stored in non-publicly available Available on request

REFERENCES:
- [Result] Ralapanawa U, Sivakanesan R. Epidemiology and the Magnitude of Coronary Artery Disease and Acute Coronary Syndrome: A Narrative Review. J Epidemiol Glob Health. 2021 Jun;11(2):169-177. doi: 10.2991/jegh.k.201217.001. Epub 2021 Jan 7. PMID 33605111
- [Result] Velilla Moliner J, Gros Baneres B, Povar Marco J, Santalo Bel M, Ordonez Llanos J, Martin Martin A, Temboury Ruiz F. Diagnostic performance of high sensitive troponin in non-ST elevation acute coronary syndrome. Med Intensiva (Engl Ed). 2020 Mar;44(2):88-95. doi: 10.1016/j.medin.2018.07.014. Epub 2018 Sep 21. English, Spanish. PMID 30249382
- [Result] Castro LT, Santos IS, Goulart AC, Pereira ADC, Staniak HL, Bittencourt MS, Lotufo PA, Bensenor IM. Elevated High-Sensitivity Troponin I in the Stabilized Phase after an Acute Coronary Syndrome Predicts All-Cause and Cardiovascular Mortality in a Highly Admixed Population: A 7-Year Cohort. Arq Bras Cardiol. 2019 Mar;112(3):230-237. doi: 10.5935/abc.20180268. Epub 2019 Jan 7. PMID 30916200
- [Result] Vogiatzis I, Dapcevic I, Datsios A, Koutsambasopoulos K, Gontopoulos A, Grigoriadis S. A Comparison of Prognostic Value of the Levels of ProBNP and Troponin T in Patients with Acute Coronary Syndrome (ACS). Med Arch. 2016 Jul 27;70(4):269-273. doi: 10.5455/medarh.2016.70.269-273. PMID 27703287
- [Result] Qin Z, Du Y, Zhou Q, Lu X, Luo L, Zhang Z, Guo N, Ge L. NT-proBNP and Major Adverse Cardiovascular Events in Patients with ST-Segment Elevation Myocardial Infarction Who Received Primary Percutaneous Coronary Intervention: A Prospective Cohort Study. Cardiol Res Pract. 2021 Nov 2;2021:9943668. doi: 10.1155/2021/9943668. eCollection 2021. PMID 34765262